CLINICAL TRIAL: NCT02230189
Title: Mechanistic Study of Epithelial miRNAs and T-cell Recruitment Dynamics That Occur After Allergen Challenge in Patients With Asthma.
Brief Title: Study of the Inflammation and Airway Changes That Occur After Exposure to Allergen in Asthmatics
Acronym: ACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prescott Woodruff (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Prescott Woodruff, Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-14224; 5U19AI077439 (NIH)
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Asthma
Keywords: Asthma; Allergen challenge
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy; Spirometry

STUDY DESIGN:
Intervention Model Description: Single group before and after administration of allergen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allergen challenge subjects (Experimental): Intervention: Segmental airway allergen challenge
  Three types of subjects are studied in this arm:
  1) Volunteers with neither asthma nor allergy (as established by skin prick testing); 2) Volunteers with allergy (as established by skin prick testing) but without asthma; and 3) Volunteers with both asthma and allergy (as established by skin prick testing)
  Interventions: Biological: Segmental airway allergen challenge; Procedure: Bronchoscopy; Diagnostic Test: Methacholine challenge test; Diagnostic Test: Spirometry; Diagnostic Test: Allergen skin prick test

INTERVENTIONS:
Biological: Segmental airway allergen challenge
Procedure: Bronchoscopy
Diagnostic Test: Methacholine challenge test
Diagnostic Test: Spirometry
Diagnostic Test: Allergen skin prick test

SUMMARY:
This protocol describes a single site mechanistic study to investigate microRNAs (miRNAs) that are differentially expressed in the airway epithelium of patients with asthma at baseline and in response to allergen challenge. We hypothesize that allergen exposure enhances airway smooth muscle contractility and epithelial cell mRNA/miRNA production as a consequence of locally increased T-cell derived cytokine production. The study will involve three visits over the course of approximately 14 days. At Visit 1, participants will be characterized in detail with lung function testing, methacholine challenge testing, and allergen skin prick testing. At Visit 2, participants will undergo bronchoscopy with segmental allergen administration of either cat or dust mite standardized allergen extract. At Visit 3 (either 24 hours later or 7 days later), bronchoscopy will be performed to collect airway samples including bronchoalveolar lavage (BAL), epithelial brushings and endobronchial biopsies. Sample analysis will include measurement of miRNA and mRNA expression in epithelial brushings (RNAseq and qPCR); analysis of cell surface markers on BAL cells and blood cells; and collection of endobronchial biopsies for immunostaining of immune cells localization, immunoblotting of smooth cell protein phosphorylation, analysis of mucin content and smooth muscle cell subculture. A total of 38 subjects (26 asthmatics with stable or well-controlled asthma, 6 allergic non-asthmatics and 6 non-allergic non-asthmatics) will complete the study.

ELIGIBILITY:
Allergic/Non-Asthmatic subjects and Allergic/Asthmatic subjects

Inclusion Criteria:

* Positive skin test to dust mite or cat allergen

Non-Allergic/Non-Asthmatic subjects

Inclusion Criteria:

* Negative skin test to panel of 12 allergens, including dust mite and cat allergen

All groups

Exclusion Criteria:

* History of intubation for asthma exacerbation
* Use of Xolair (omalizumab) within the last 6 months
* Immunotherapy with cat or dust mite extract now or in the past 5 years
* ≥ 10 pack-years smoking or any smoking in the past year
* Other lung diseases, such as sarcoidosis, bronchiectasis or active lung infection
* History of dermatographia
* History of anaphylaxis to cat allergen
* Participation in another research study involving a drug or biologic during the past 30 days
* Presence of past or current medical problems/other factors that may pose additional risks from participation or influence study results, as determined per study investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prescott G Woodruff, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Airway Clinical Research Center — http://acrc.ucsf.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Allergic Asthmatics(AA): Volunteers with both asthma and allergy (as established by skin prick testing)
- Allergic Non-Asthmatics(ANA): Volunteers with allergy (as established by skin prick testing) but without asthma;
- Non-Allergic Non-Asthmatics(NANA): Volunteers with neither asthma nor allergy (as established by skin prick testing)
Period: Overall Study
Arm/Group | Allergic Asthmatics(AA) | Allergic Non-Asthmatics(ANA) | Non-Allergic Non-Asthmatics(NANA)
Started | 22 | 2 | 4
Completed | 17 | 2 | 3
Not Completed | 5 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Allergic Non-asthmatics(ANA): ) Volunteers with allergy (as established by skin prick testing) but without asthma
- Total: Total of all reporting groups
Arm/Group | Allergic Non-asthmatics(ANA) | Non-allergic Non-asthmatics(NANA) | Allergic Asthmatics(AA) | Total
Number analyzed (Participants) | 2 | 3 | 17 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 2 | 3 | 16 | 21
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (2.12) | 29 (5) | 29.7 (7.15) | 29.5 (9.268)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 11 | 13
  Male | 1 | 2 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 4 | 5
  Not Hispanic or Latino | 1 | 3 | 13 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 2 | 3
  White | 2 | 1 | 8 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 17 | 22
FEV1 [Mean (Standard Deviation); unit: liters] | 4.52 (1.71) | 4.22 (0.397) | 3.38 (0.789) | 3.6 (0.864)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Expression of Epithelial miRNAs (in Read Counts) 24 Hours After Allergen-challenge as Compared to 24 Hours After Diluent Challenge in Participants With Allergic Asthma
Description: For each participant with Allergic Asthma, a baseline airway epithelial brushing was performed, allergen was instilled into one segment of the lung, and diluent (control) was instilled into another segment. Both segments were brushed for epithelial cells 24 hours later. After processing brushes to RNA and generating RNA sequencing data, the RNA transcript read counts for each gene underwent variance stabilized log normalization. Then we built a regression model which estimated the difference in miRNA read count in the allergen challenged as compared to the baseline sample and the difference in miRNA read count in the diluent challenged segment as compared to baseline for each participant. The change from baseline read count for each miRNA in the allergen samples was compared to the change in the diluent samples and statistical significance was assessed using the unadjusted p-value(<0.05). The direction of change does not have clinical significance; this was a mechanistic study.
Time Frame: 24 hours
Population: Our pre-specified primary outcome was limited to Allergic Asthmatics only. The rationale for this is that participants without allergy or asthma do not respond to Allergen Challenge and therefore the changes in miRNA are uninformative.
Measure: Mean (Standard Deviation); unit: Normalized log2 copy number
Groups:
- Allergen Challenge Subjects: Intervention: Segmental airway allergen challenge
  In this arm, we studied volunteers with both asthma and allergy (as established by skin prick testing)
  Biological/Vaccine: Segmental airway allergen challenge Procedure/Surgery: Bronchoscopy Diagnostic Test: Methacholine challenge test Diagnostic Test: Spirometry Diagnostic Test: Allergen skin prick test
- Diluent Challenge Subjects: Intervention: Segmental airway diluent challenge
  In this arm, we studied volunteers with both asthma and allergy (as established by skin prick testing).
Arm/Group | Allergen Challenge Subjects | Diluent Challenge Subjects
Number analyzed (Participants) | 12 | 12
Normalized log2 copy number
  miR4521 | 7.33 (0.79) | 6.74 (0.43)
  miR107 | 9.63 (0.61) | 9.01 (0.98)
  miR891a | 7.02 (0.64) | 6.56 (0.46)
  miR363 | 9.55 (1.16) | 8.77 (1.07)
  miR1248 | 7.02 (0.31) | 7.21 (0.48)
  miR944 | 7.12 (0.19) | 7.27 (0.36)
  miR6806 | 6.63 (0.22) | 6.35 (0.13)
  miR103a | 12.05 (0.38) | 11.7 (0.48)
  miR454-5p | 6.77 (0.16) | 6.57 (0.28)
  miR320e | 6.57 (0.16) | 6.69 (0.24)
  miR181a | 8.29 (0.33) | 8.83 (0.86)
  miR130b | 6.72 (0.17) | 6.5 (0.33)
  miR365a | 6.4 (0.14) | 6.55 (0.21)
  miR135b | 6.65 (0.22) | 6.43 (0.19)
  miR1273h | 6.53 (0.24) | 6.62 (0.33)
  miR3177 | 6.79 (0.26) | 6.88 (0.27)
Statistical Analysis 1: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR4521; Test type: Superiority; p = 0.010, t-test, 2 sided; Mean Difference (Net) = 2.11
Statistical Analysis 2: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR107; Test type: Superiority; p = 0.010, t-test, 2 sided; Mean Difference (Net) = 0.56
Statistical Analysis 3: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR-891a; Test type: Superiority; p = 0.018, t-test, 2 sided; Mean Difference (Net) = 2.57
Statistical Analysis 4: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR363; Test type: Superiority; p = 0.021, t-test, 2 sided; Mean Difference (Net) = 0.88
Statistical Analysis 5: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR1248; Test type: Superiority; p = 0.028, t-test, 2 sided; Mean Difference (Net) = -1
Statistical Analysis 6: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR944; Test type: Superiority; p = 0.033, t-test, 2 sided; Mean Difference (Net) = -0.85
Statistical Analysis 7: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR6806; Test type: Superiority; p = 0.034, t-test, 2 sided; Mean Difference (Net) = 2.13
Statistical Analysis 8: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR103a; Test type: Superiority; p = 0.036, t-test, 2 sided; Mean Difference (Net) = 0.39
Statistical Analysis 9: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR454; Test type: Superiority; p = 0.037, t-test, 2 sided; Mean Difference (Net) = 1.69
Statistical Analysis 10: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR320e; Test type: Superiority; p = 0.041, t-test, 2 sided; Mean Difference (Net) = -1.13
Statistical Analysis 11: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR181a; Test type: Superiority; p = 0.043, t-test, 2 sided; Mean Difference (Net) = -0.55
Statistical Analysis 12: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR130b; Test type: Superiority; p = 0.044, t-test, 2 sided; Mean Difference (Net) = 1.95
Statistical Analysis 13: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR365a; Test type: Superiority; p = 0.044, t-test, 2 sided; Mean Difference (Net) = -2.18
Statistical Analysis 14: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR135b; Test type: Superiority; p = 0.047, t-test, 2 sided; Mean Difference (Net) = 2.06
Statistical Analysis 15: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR1273h; Test type: Superiority; p = 0.048, t-test, 2 sided; Mean Difference (Net) = -2.35
Statistical Analysis 16: Comparison: Allergen Challenge Subjects vs Diluent Challenge Subjects; miR3177; Test type: Superiority; p = 0.048, t-test, 2 sided; Mean Difference (Net) = -1.31

2. Primary Outcome: Difference in Expression of Epithelial miRNAs (in Read Counts) 7 Days After Allergen-challenge as Compared to 7 Days After Diluent Challenge
Description: For each participant with Allergic Asthma, a baseline airway epithelial brushing was performed, allergen was instilled into one segment of the lung, and diluent (control) was instilled into another segment. Both segments were brushed for epithelial cells 7 days later. After processing the brushes to RNA and generating RNA sequencing data, the RNA transcript read counts for each gene underwent variance stabilized log normalization. Then we built a regression model which estimated the difference in miRNA read count in the allergen challenged as compared to the baseline sample and the difference in miRNA read count in the diluent challenged segment as compared to baseline for each participant. The change from baseline read count for each miRNA in the allergen samples was compared to the change in the diluent samples and statistical significance was assessed using the unadjusted p-value(<0.05). The direction of change does not have clinical significance; this was a mechanistic study.
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Normalized log2 copy number
Groups:
- Allergen Challenge Segment: Intervention: Segmental airway allergen challenge
  In this arm, we studied volunteers with both asthma and allergy (as established by skin prick testing)
  Biological/Vaccine: Segmental airway allergen challenge Procedure/Surgery: Bronchoscopy Diagnostic Test: Methacholine challenge test Diagnostic Test: Spirometry Diagnostic Test: Allergen skin prick test
- Diluent Challenge Segment: Intervention: Segmental airway diluent challenge
  In this arm, we studied volunteers with both asthma and allergy (as established by skin prick testing).
Arm/Group | Allergen Challenge Segment | Diluent Challenge Segment
Number analyzed (Participants) | 4 | 4
Normalized log2 copy number
  miR6510 | 7.74 (0.57) | 9.2 (0.81)
  miR3605 | 5.92 (0.61) | 6.9 (0.8)
  miR3912 | 5.03 (0.53) | 5.83 (0.61)
  miR15b | 6.76 (0.33) | 6.09 (0.39)
  miR127 | 7.06 (0.8) | 8.54 (1.73)
  miR146a | 14.14 (1.19) | 12.73 (0.8)
  miR449b | 9.99 (0.54) | 8.84 (0.88)
  miR21-5p | 18.02 (0.33) | 17 (0.82)
  miR6842 | 6.83 (0.37) | 7.67 (0.44)
  miR142-5p | 7.68 (0.38) | 6.93 (0.66)
  miR21 | 7.97 (0.49) | 6.83 (0.99)
  miR493 | 5.03 (0.31) | 5.66 (0.67)
  miR193a | 6.66 (0.99) | 7.46 (0.72)
  miR149 | 9.98 (0.42) | 10.95 (0.4)
  miR449a | 12.46 (0.56) | 11.36 (0.95)
  miR6511a | 5.58 (0.66) | 6.46 (0.56)
  miR6843 | 5.99 (0.11) | 6.8 (0.67)
  miR671 | 8.53 (0.87) | 9.3 (0.73)
  miR6503 | 4.93 (0.19) | 5.56 (0.59)
  miR450b | 6.05 (0.4) | 5.35 (0.52)
  miR485 | 5.08 (0.62) | 5.68 (0.72)
  miR6806 | 5.22 (0.38) | 5.85 (0.43)
  miR3182 | 5.92 (0.2) | 5.68 (0.97)
  miR142-3p | 7.58 (0.21) | 6.72 (0.91)
  miR320d | 6.48 (0.33) | 7.09 (0.72)
  miR3928 | 5.95 (0.3) | 5.24 (0.49)
  miR744 | 5.6 (0.58) | 5.1 (0.47)
  miR206 | 5.67 (1.06) | 5.18 (0.61)
  miR30e | 11.3 (0.29) | 10.36 (0.7)
  miR4500 | 6.21 (0.41) | 5.61 (0.22)
  miR125a | 13.66 (1.47) | 14.55 (1.18)
  miR99b | 13.78 (0.31) | 14.33 (0.4)
  miR1 | 5.86 (0.76) | 5.17 (0.49)
  miR146b | 14.13 (0.38) | 14.72 (0.76)
  miR1255a | 5.21 (0.54) | 5.79 (0.67)
  miR223 | 9.9 (0.6) | 8.9 (1.08)
  miR642a | 7.8 (0.56) | 8.32 (0.22)
  miR548ae | 5.86 (0.24) | 5.23 (0.4)
  miR146b-3p | 7.9 (0.35) | 8.58 (0.31)
  miR877 | 5.13 (0.42) | 5.66 (0.39)
  miR181a | 8.25 (0.32) | 8.74 (0.58)
  miR4467 | 5.17 (0.47) | 5.56 (0.92)
  miR1249 | 5.05 (0.35) | 5.62 (0.44)
  miR766 | 5.59 (0.63) | 4.98 (0.3)
  miR29c | 7.93 (0.56) | 7.09 (0.78)
  miR370 | 5.77 (0.76) | 6.51 (1)
Statistical Analysis 1: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR6510; Test type: Superiority; p = 0.0, t-test, 2 sided; Mean Difference (Net) = -1.83
Statistical Analysis 2: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR3605; Test type: Superiority; p = 0, t-test, 2 sided; Mean Difference (Net) = -2.09
Statistical Analysis 3: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR3912; Test type: Superiority; p = 0, t-test, 2 sided; Mean Difference (Net) = -5.75
Statistical Analysis 4: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR15b; Test type: Superiority; p = 0, t-test, 2 sided; Median Difference (Net) = 1.93
Statistical Analysis 5: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR127; Test type: Superiority; p = 0, t-test, 2 sided; Mean Difference (Net) = -2.35
Statistical Analysis 6: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR146a; Test type: Superiority; p = 0, t-test, 2 sided; Mean Difference (Net) = 1.59
Statistical Analysis 7: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR449b; Test type: Superiority; p = 0, t-test, 2 sided; Mean Difference (Net) = 1.21
Statistical Analysis 8: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR21-5p; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 0.85
Statistical Analysis 9: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR6842; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -1.29
Statistical Analysis 10: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR142-5p; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 1.24
Statistical Analysis 11: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR21; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 1.67
Statistical Analysis 12: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR493; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -4.24
Statistical Analysis 13: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR193a; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -1.46
Statistical Analysis 14: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR149; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -0.89
Statistical Analysis 15: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR449a; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 1.06
Statistical Analysis 16: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR6511a; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -2.1
Statistical Analysis 17: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR6843; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -1.59
Statistical Analysis 18: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR671; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Net) = -0.95
Statistical Analysis 19: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR6503; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -4.65
Statistical Analysis 20: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR450b; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = 2.84
Statistical Analysis 21: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR485; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -4.92
Statistical Analysis 22: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR6806; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -2.49
Statistical Analysis 23: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR3182; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = 2.18
Statistical Analysis 24: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR142-3p; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = 1.28
Statistical Analysis 25: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR320d; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -1.23
Statistical Analysis 26: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR3928; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = 2.73
Statistical Analysis 27: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR744; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = 4.59
Statistical Analysis 28: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR206; Test type: Superiority; p = 0.02, t-test, 2 sided; Median Difference (Net) = 3.42
Statistical Analysis 29: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR30e; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = 0.9
Statistical Analysis 30: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR4500; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = 1.52
Statistical Analysis 31: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR125a; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = -0.98
Statistical Analysis 32: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR99b; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = -0.6
Statistical Analysis 33: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR1; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = 2.67
Statistical Analysis 34: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR146b; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = -0.77
Statistical Analysis 35: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR1255a; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = -3.17
Statistical Analysis 36: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR223; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = 1.02
Statistical Analysis 37: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR642a; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Net) = -0.78
Statistical Analysis 38: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR548ae; Test type: Superiority; p = 0.4, t-test, 2 sided; Mean Difference (Net) = 2.17
Statistical Analysis 39: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR146b; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Net) = -0.79
Statistical Analysis 40: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR877; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Net) = -2.52
Statistical Analysis 41: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR181a; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Net) = -0.69
Statistical Analysis 42: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR4467; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Net) = -3.4
Statistical Analysis 43: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR1249; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Net) = -2.48
Statistical Analysis 44: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR766; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Net) = 3.87
Statistical Analysis 45: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR29c; Test type: Superiority; p = 0.048, t-test, 2 sided; Mean Difference (Net) = 1.07
Statistical Analysis 46: Comparison: Allergen Challenge Segment vs Diluent Challenge Segment; miR370; Test type: Superiority; p = -1.75, t-test, 2 sided; Mean Difference (Net) = -1.75

ADVERSE EVENTS:
Time Frame: Adverse event data were prospectively collected from the first visit until 48 hours after the last study visit in all participants and until the resolution of any potential adverse event reported by a subject after a study procedure, up to 6 months.
Arm/Group | Allergic Asthmatics(AA) | Allergic Non-Asthmatics(ANA) | Non-Allergic Non-Asthmatics(NANA)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/22 | 0/2 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allergic Asthmatics(AA) (N=22) | Allergic Non-Asthmatics(ANA) (N=2) | Non-Allergic Non-Asthmatics(NANA) (N=4)
Pregnancy identified during study enrollment (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — Participant was not pregnant upon enrollment (confirmed via urine pregnancy test). Participant later notified study team of pregnancy and was withdrawn prior to Visit 2 and Visit 3 bronchoscopies. Event was reported to sponsor and medical monitor.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allergic Asthmatics(AA) (N=22) | Allergic Non-Asthmatics(ANA) (N=2) | Non-Allergic Non-Asthmatics(NANA) (N=4)
Increased systolic blood pressure post-bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory infection post-bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT02230189/Prot_SAP_000.pdf